CLINICAL TRIAL: NCT01229475
Title: Stepwise Approach Versus Linear Ablation for Repeat Procedure in Patients With Recurrence of Persistent Atrial Fibrillation
Brief Title: Stepwise Approach Versus Linear Ablation in Patients With Recurrence of Persistent Atrial Fibrillation
Acronym: REDO-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Isabel Deisenhofer, MD and Sonia Ammar, MD, Deutsches Herzzentrum München
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-003
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation; Recurrence
Keywords: Atrial fibrillation; recurrence; repeat procedure; linear ablation; stepwise approach
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepwise approach (Active Comparator): Stepwise approach for repeat AF ablation
  Interventions: Procedure: Ablation with stepwise approach; Procedure: Linear ablation
- Linear ablation (Active Comparator): Linear ablation for repeat procedure in patients with recurrent atrial fibrillation
  Interventions: Procedure: Ablation with stepwise approach; Procedure: Linear ablation

INTERVENTIONS:
Procedure: Ablation with stepwise approach — Stepwise approach for repeat AF ablation
Procedure: Linear ablation — Linear ablation for AF ablation

SUMMARY:
Catheter ablation of persistent atrial fibrillation (AF) remains a challenging procedure. Even in experienced centres, repeat interventions are necessary in up to 70 of patients to achieve sinus rhythm at a long-term follow-up.

While there is a consensus to perform pulmonary vein isolation (PVI) as a cornerstone for the ablation of paroxysmal and persistent AF ablation, different additional ablation strategies are used to achieve a modification of the substrate that perpetuates the arrhythmia: linear lesions (anterior and roof lines) or ablation of complex fractionated atrial electrograms (CFAE). In the stepwise approach PVI, CFAE ablation and/or LL are combined according to the presenting arrhythmia during procedure.

The aim of the study is to determine whether there is a difference in terms of freedom from arrhythmia between a stepwise approach and a linear ablation for repeat procedure in patient with recurrence of persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrence of symptomatic persistent atrial fibrillation after at least one ablation procedure,
* with the last ablation procedure at least 3 months ago.
* at least one unsuccessful attempt of antiarrhythmic drug
* oral anticoagulation for at least 4 weeks prior to ablation

Exclusion Criteria:

* LA thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia
  Documented freedom from atrial arrhythmia (AF or AT) during follow-up.

SECONDARY OUTCOMES:
Procedural and safety data
  1. Duration of left atrial procedure, ablation time, fluoroscopy time.
  2. Complications
  3. Type of recurrent arrhythmia
  4. Number of reablation

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum München; Sonia Ammar, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Germany